CLINICAL TRIAL: NCT01634191
Title: An Open-Label, Single-Dose Study to Evaluate the Effects of Age and Sex on the Pharmacokinetics of Apremilast (CC-10004) in Healthy Subjects
Brief Title: Effects of Age and Sex on the Pharmacokinetics of Apremilast in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CC-10004-CP-024; 20200149 (Other: Amgen Study ID)
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteer
Keywords: Apremilast; pharmacokinetic; safety; Pharmacokinetics and safety in healthy volunteer subjects
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elderly: Apremilast 30 mg (Experimental): Participants aged 65 to 85 years received a single oral dose of 30 mg apremilast on Day 1.
  Interventions: Drug: Apremilast
- Younger: Apremilast 30 mg (Experimental): Participants aged 18 to 55 years received a single oral dose of 30 mg apremilast on Day 1.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — One oral 30 mg dose of apremilast
  Other Names: CC-10004; Otezla®

SUMMARY:
The purpose of the study is to evaluate the effects of age and sex on the pharmacokinetics and safety of a single oral dose of 30 mg apremilast in healthy adults.

DETAILED DESCRIPTION:
This is an open-label, parallel group study where eligible elderly adults (aged 65-85 years inclusive) and younger adults (aged 18-55 years inclusive) and who are matched to the elderly participants by sex and body mass index (BMI) (± 10%) will receive a single dose of 30 mg apremilast under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for elderly group

1. Healthy male or female subjects of any ethnic origin between ages of 65 and 85 inclusive with a body mass index (BMI) between 18 and 35.
2. Females must have been surgically sterilized at least 6 months prior to screening or be postmenopausal (to be confirmed by lab tests).
3. Males must agree to use latex or polyurethane condoms when engaging in sex during the study and for at least 28 days after dosing.
4. Elderly subjects with stable, chronic medical condition may be eligible if the condition is well-controlled and medications do not interfere with study procedures or pharmacokinetic interpretation

Inclusion Criteria for younger group:

1. Healthy male or female of any ethnic origin between the ages of 18 and 55 inclusive with a BMI between 18 and 35.
2. Males must agree to use latex or polyurethane condoms when engaging in sex during the study and for at least 28 days after dosing.
3. Females who are able to become pregnant have a negative pregnancy test at screening and baseline, and must agree to use one of the following:

   * a highly effective form of contraception (ex. Non-oral hormonal, intrauterine device) OR
   * oral hormonal contraceptive plus one additional form of barrier contraception OR
   * two forms of barrier contraception These must be effective by the time of screening. For younger females who are not able to become pregnant, the conditions for the elderly females will apply.

Exclusion Criteria:

1. Any condition, including the presence of laboratory abnormalities, or psychiatric illness, that would prevent the subject from signing the Informed Consent form, places the subject at unacceptable risk if he were to participate in the study, or confounds the ability to interpret data from the study.
2. Presence of any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, and excretion, or plans to have elective or medical procedures during the conduct of the trial.
3. Exposure to an investigational drug (new chemical entity) within 30 days prior to the first dose administration or 5 half-lives of that investigational drug, if known (whichever is longer).
4. Subjects with known serum hepatitis, is a known carrier of hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus antibody.
5. Subjects who have used prescription systemic or topical medications within 30 days of dosing, unless it is being used to treat a stable, chronic medical condition. This includes medication that is an inhibitor or inducer of P-glycoprotein transporter and CYP-3A4/5 used within 14 days of dosing.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2012-03-01 (Actual); Study Completion 2012-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - PRA International, Lenexa, Kansas
  - Clinical Development Services, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at two clinical research sites in the United States.
Groups:
- Young: Apremilast 30 mg: Participants aged 18 to 55 years received a single oral dose of 30 mg apremilast on Day 1.
Period: Overall Study
Arm/Group | Young: Apremilast 30 mg | Elderly: Apremilast 30 mg
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Young Males: Men aged 18 to 55 years received a single oral dose of 30 mg apremilast on Day 1.
- Young Females: Women aged 18 to 55 years received a single oral dose of 30 mg apremilast on Day 1.
- Elderly Males: Men aged 65 to 85 years received a single oral dose of 30 mg apremilast on Day 1.
- Elderly Females: Women aged 65 to 85 years received a single oral dose of 30 mg apremilast on Day 1.
- Total: Total of all reporting groups
Arm/Group | Young Males | Young Females | Elderly Males | Elderly Females | Total
Number analyzed (Participants) | 8 | 10 | 8 | 10 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (7.48) | 35.2 (7.19) | 70.4 (3.62) | 70.6 (4.72) | 52.4 (19.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 10 | 0 | 10 | 20
  Male | 8 | 0 | 8 | 0 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 8 | 8 | 8 | 10 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 4 | 8 | 8 | 24
  Black or African American | 3 | 6 | 0 | 2 | 11
  Other | 1 | 0 | 0 | 0 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.6 (2.43) | 27.5 (2.59) | 26.3 (2.69) | 27.1 (2.42) | 26.9 (2.47)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC0-t) of Apremilast
Description: The lower limit of quantitation for apremilast plasma concentrations was 1.0 ng/mL.
  AUC0-t was calculated using the linear trapezoidal method when concentrations were increasing and the logarithmic trapezoidal method when concentrations were decreasing.
Time Frame: Day 1 predose and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The pharmacokinetic (PK) population included all participants who received apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Young: Apremilast: Participants aged 18 to 55 years received a single oral dose of 30 mg apremilast on Day 1.
- Elderly: Apremilast: Participants aged 65 to 85 years received a single oral dose of 30 mg apremilast on Day 1.
Arm/Group | Young: Apremilast | Elderly: Apremilast
Number analyzed (Participants) | 18 | 18
h*ng/mL | 2832 (28.1) | 3235 (40.3)
Statistical Analysis 1: Comparison: Young: Apremilast vs Elderly: Apremilast; To assess the effect of age on the PK of apremilast after a single 30 mg dose, a 2-way analysis of variance (ANOVA) model was performed on the log-transformed AUC0-t. The ANOVA model included age group (elderly and young), sex (male and female), and age group by sex as a fixed effect; Test type: Other; Geometric Mean Ratio = 113, 90% CI 2-sided [94.2 to 135] — Geometric mean ratio (Elderly/Young) and 90% confidence interval (CI) of the ratio calculated from a 2-way ANOVA model, and presented as percentages

2. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) was any noxious, unintended, or untoward medical occurrence that appeared or worsened in a participant during the course of the study. It could have been a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health including laboratory test values, regardless of etiology. Any worsening (i.e., any clinically significant adverse change in the frequency or intensity of a pre-existing condition) was considered an AE.
Time Frame: From first dose of study drug up to 11 days
Population: Participants who received apremilast
Measure: Count of Participants; unit: Participants
Arm/Group | Young Males | Young Females | Elderly Males | Elderly Females
Number analyzed (Participants) | 8 | 10 | 8 | 10
Participants
  Any adverse event | 2 | 1 | 2 | 5
  Adverse event related to study drug | 2 | 1 | 0 | 1
  Serious adverse events | 0 | 0 | 0 | 0
  Serious adverse events related to study drug | 0 | 0 | 0 | 0
  Discontinued due to adverse event | 0 | 0 | 0 | 0
  Discontinued due to adverse event related to study drug | 0 | 0 | 0 | 0

3. Primary Outcome: AUC From Time Zero to Time of Last Quantifiable Concentration (AUC0-t) of Apremilast by Sex
Description: as for outcome 1
Time Frame: Day 1 predose and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Males (Combined): Male participants received a single oral dose of 30 mg apremilast on Day 1.
- Females (Combined): Female participants received a single oral dose of 30 mg apremilast on Day 1.
Arm/Group | Males (Combined) | Females (Combined)
Number analyzed (Participants) | 16 | 20
h*ng/mL | 2634 (24.5) | 3382 (38.2)
Statistical Analysis 1: Comparison: Males (Combined) vs Females (Combined); To assess the effect of sex on the PK of apremilast after a single 30 mg dose, a 2-way analysis of variance (ANOVA) model was performed on the log-transformed AUC0-t. The ANOVA model included age group (elderly and young), sex (male and female), and age group by sex as a fixed effect; Test type: Other; Geometric Mean Ratio = 128, 90% CI 2-sided [107 to 154] — Geometric mean ratio (Female/Male) and 90% CI of the ratio calculated from a 2-way ANOVA model, and presented as percentages

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-∞) of Apremilast
Description: The lower limit of quantitation for apremilast plasma concentrations was 1.0 ng/mL.
Time Frame: Day 1 predose and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Young: Apremilast | Elderly: Apremilast
Number analyzed (Participants) | 18 | 18
h*ng/mL | 2900 (28.7) | 3323 (41.8)
Statistical Analysis 1: Comparison: Young: Apremilast vs Elderly: Apremilast; To assess the effect of age on the PK of apremilast after a single 30 mg dose, a 2-way analysis of variance (ANOVA) model was performed on the log-transformed AUC0-∞. The ANOVA model included age group (elderly and young), sex (male and female), and age group by sex as a fixed effect; Test type: Other; Geometric Mean Ratio = 113, 90% CI 2-sided [94.1 to 135] — Geometric mean ratio (Elderly/Young) and 90% CI of the ratio calculated from a 2-way ANOVA model, and presented as percentages

5. Primary Outcome: AUC From Time Zero Extrapolated to Infinity (AUC0-∞) of Apremilast by Sex
Description: The lower limit of quantitation for apremilast plasma concentrations was 1.0 ng/mL.
Time Frame: Day 1 predose and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Males (Combined) | Females (Combined)
Number analyzed (Participants) | 16 | 20
h*ng/mL | 2673 (24.8) | 3499 (39.1)
Statistical Analysis 1: Comparison: Males (Combined) vs Females (Combined); To assess the effect of sex on the PK of apremilast after a single 30 mg dose, a 2-way ANOVA model was performed on the log-transformed AUC0-∞. The ANOVA model included age group (elderly and young), sex (male and female), and age group by sex as a fixed effect; Test type: Other; Geometric Mean Ratio = 131, 90% CI 2-sided [109 to 157] — [estimate comment as in outcome 3, analysis 1]

6. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Apremilast
Description: The lower limit of quantitation for apremilast plasma concentrations was 1.0 ng/mL.
Time Frame: Day 1 predose and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Young: Apremilast | Elderly: Apremilast
Number analyzed (Participants) | 18 | 18
ng/mL | 302 (26.8) | 321 (27.8)
Statistical Analysis 1: Comparison: Young: Apremilast vs Elderly: Apremilast; To assess the effect of age on the PK of apremilast after a single 30 mg dose, a 2-way analysis of ANOVA model was performed on the log-transformed Cmax. The ANOVA model included age group (elderly and young), sex (male and female), and age group by sex as a fixed effect; Test type: Other; Geometric Mean Ratio = 106, 90% CI 2-sided [90.5 to 123] — [estimate comment as in outcome 4, analysis 1]

7. Primary Outcome: Maximum Observed Plasma Concentration of Apremilast by Sex
Description: The lower limit of quantitation for apremilast plasma concentrations was 1.0 ng/mL.
Time Frame: Day 1 predose and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Males (Combined) | Females (Combined)
Number analyzed (Participants) | 16 | 20
ng/mL | 299 (16.6) | 322 (33.5)
Statistical Analysis 1: Comparison: Males (Combined) vs Females (Combined); To assess the effect of sex on the PK of apremilast after a single 30 mg dose, a 2-way ANOVA model was performed on the log-transformed Cmax. The ANOVA model included age group (elderly and young), sex (male and female), and age group by sex as a fixed effect; Test type: Other; Geometric Mean Ratio = 108, 90% CI 2-sided [92.3 to 126] — [estimate comment as in outcome 3, analysis 1]

8. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Apremilast
Description: The lower limit of quantitation for apremilast plasma concentrations was 1.0 ng/mL.
Time Frame: Day 1 predose and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received apremilast and had evaluable PK profiles.
Measure: Median (Full Range); unit: hours
Arm/Group | Young: Apremilast | Elderly: Apremilast
Number analyzed (Participants) | 18 | 18
hours | 2.50 [0.5 to 5.0] | 2.50 [1.0 to 5.1]
Statistical Analysis 1: Comparison: Young: Apremilast vs Elderly: Apremilast; Tmax was analyzed by nonparametric methods. The median difference and 90% CI of the median difference were calculated from the Hodges-Lehrmann estimate; Test type: Other; p = 0.153, Wilcoxon rank-sum test; Median Difference = 0.500, 90% CI 2-sided [0.000 to 2.00] — Median difference (Elderly - Young) calculated from the Hodges-Lehmann estimate

9. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Apremilast by Sex
Description: The lower limit of quantitation for apremilast plasma concentrations was 1.0 ng/mL.
Time Frame: Day 1 predose and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received apremilast and had evaluable PK profiles.
Measure: Median (Full Range); unit: hours
Arm/Group | Males (Combined) | Females (Combined)
Number analyzed (Participants) | 16 | 20
hours | 2.5 [0.5 to 5.0] | 2.75 [1.0 to 5.1]
Statistical Analysis 1: Comparison: Males (Combined) vs Females (Combined); [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.169, Wilcoxon rank-sum test; Median Difference = 0.500, 90% CI 2-sided [0.000 to 2.00] — Median difference (Female - Male) and 90% CI of the difference calculated from the Hodges-Lehmann estimate

10. Primary Outcome: Estimate of Terminal Elimination Half-life of Apremilast in Plasma (t1/2)
Time Frame: Day 1 predose and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received apremilast and had evaluable PK profiles.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Young: Apremilast | Elderly: Apremilast
Number analyzed (Participants) | 18 | 18
hours | 9.41 (2.65) | 9.15 (2.56)

11. Primary Outcome: Estimate of Terminal Elimination Half-life of Apremilast in Plasma by Sex
Time Frame: Day 1 predose and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received apremilast and had evaluable PK profiles.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Males (Combined) | Females (Combined)
Number analyzed (Participants) | 16 | 20
hours | 8.06 (1.72) | 10.3 (2.76)

12. Primary Outcome: Apparent Total Plasma Clearance When Dosed Orally (CL/F) of Apremilast
Time Frame: Day 1 predose and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Young: Apremilast | Elderly: Apremilast
Number analyzed (Participants) | 18 | 18
L/hr | 10.4 (28.7) | 9.03 (41.8)

13. Primary Outcome: Apparent Total Plasma Clearance When Dosed Orally of Apremilast by Sex
Time Frame: Day 1 predose and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Males (Combined) | Females (Combined)
Number analyzed (Participants) | 16 | 20
L/hr | 11.2 (24.8) | 8.57 (39.1)

14. Primary Outcome: Apparent Total Volume of Distribution When Dosed Orally (Vz/F) of Apremilast
Time Frame: Day 1 predose and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Young: Apremilast | Elderly: Apremilast
Number analyzed (Participants) | 18 | 18
liters | 136 (38.9) | 115 (35.3)

15. Primary Outcome: Apparent Total Volume of Distribution When Dosed Orally (Vz/F) of Apremilast by Sex
Time Frame: Day 1 predose and at 0.5, 1, 1.5, 2, 2.5, 3, 5, 8, 12, 24, 36, and 48 hours after dosing.
Population: The PK population included all participants who received apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Males (Combined) | Females (Combined)
Number analyzed (Participants) | 16 | 20
liters | 128 (30.7) | 123 (43.4)

ADVERSE EVENTS:
Time Frame: From first dose of apremilast up to 11 days
Groups:
- Young (Total): Participants aged 18 to 55 years received a single oral dose of 30 mg apremilast on Day 1.
- Elderly (Total): Participants aged 65 to 85 years received a single oral dose of 30 mg apremilast on Day 1.
- Overall Total: All study participants received a single oral dose of 30 mg apremilast on Day 1.
Arm/Group | Young Males | Young Females | Young (Total) | Elderly Males | Elderly Females | Elderly (Total) | Overall Total
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/18 | 0/8 | 0/10 | 0/18 | 0/36
Other Adverse Events (participants affected / at risk) | 2/8 | 1/10 | 3/18 | 2/8 | 5/10 | 7/18 | 10/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Young Males (N=8) | Young Females (N=10) | Young (Total) (N=18) | Elderly Males (N=8) | Elderly Females (N=10) | Elderly (Total) (N=18) | Overall Total (N=36)
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 2
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
PAIN (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
HEADACHE (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
SOMNOLENCE (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
PHLEBITIS (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.